CLINICAL TRIAL: NCT00844051
Title: Prospective Study of School-based Influenza Vaccination's Impact on School Populations
Brief Title: Study to Evaluate Impact of School-based Influenza Vaccination on School Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Pia S. Pannaraj, Assistant Professor of Pediatrics, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHLA-08-00229
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2016-08-01 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Influenza; influenza vaccination; school-based vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention (No Intervention): No school-based influenza vaccination program
- Intervention (Active Comparator): School-based Influenza Vaccination Program
  Interventions: Biological: School-based influenza vaccination program

INTERVENTIONS:
Biological: School-based influenza vaccination program — School-based influenza vaccination program
  Arms: Intervention

SUMMARY:
Rates of confirmed influenza illness in vaccinated and non-vaccinated children will be compared between schools with and without vaccination programs. The investigators hypothesize that in addition to lowering rates of influenza in vaccinated children, raising vaccination rates by 30-40% through school-based vaccination programs will decrease incidence of influenza in non-vaccinated children attending those schools compared to non-vaccinated children in schools with low vaccination rates.

DETAILED DESCRIPTION:
This prospective cohort study will evaluate rates of virologically confirmed influenza in children attending schools with and without school-based vaccination programs. Eight schools (4455 students) in two school districts matched for size, race/ethnicity, socioeconomic status, and location will serve as intervention and control schools. During influenza season defined by local surveillance data, nasal/throat swabs will be obtained for rapid influenza detection assays from all children with fever and respiratory symptoms identified by teachers for evaluation in the school nurse's office. Absent children will be offered testing at a central location within the schools' communities.Rates of confirmed influenza illness in vaccinated and non-vaccinated children will be compared between schools with and without vaccination programs. Rates of absenteeism also will be evaluated. The investigators hypothesize that in addition to lowering rates of influenza in vaccinated children, raising vaccination rates by 30-40% through school-based vaccination programs will decrease incidence of influenza in non-vaccinated children attending those schools compared to non-vaccinated children in schools with low vaccination rates.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in target schools

Exclusion Criteria: none

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4455 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia S Pannaraj, MD, MPH, Principal Investigator — Childrens Hospital Los Angeles, University of Southern California
Locations (2):
- United States (2):
  - Los Angeles County Department of Public Health, Los Angeles, California
  - Childrens Hospital Los Angeles, Los Angeles, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Intervention | Intervention
Started | 2087 | 2368
Completed | 2087 | 2368
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention | Intervention | Total
Number analyzed (Participants) | 2087 | 2368 | 4455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2087 | 2368 | 4455
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.2 [5 to 13] | 8.3 [5 to 13] | 8.3 [5 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 987 | 1146 | 2133
  Male | 1100 | 1222 | 2322
Region of Enrollment [Number; unit: participants]
  United States | 2087 | 2368 | 4455

OUTCOME MEASURES:

1. Primary Outcome: Rates of Confirmed Influenza Illness in Vaccinated and Non-vaccinated Children Attending Schools With and Without School-based Influenza Vaccination Programs
Time Frame: 1 year
Measure: Number; unit: flu+ per 1000 children
Arm/Group | No Intervention | Intervention
Number analyzed (Participants) | 2087 | 2368
flu+ per 1000 children | 58.0 | 40.1

2. Secondary Outcome: Rates of Absenteeism Among Children Attending Schools With and Without School-based Influenza Vaccination Programs
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: days per 100 school days
Arm/Group | No Intervention | Intervention
Number analyzed (Participants) | 2087 | 2368
days per 100 school days | 4.2 (4.7) | 3.9 (4.8)

ADVERSE EVENTS:
Arm/Group | No Intervention | Intervention
Serious Adverse Events (participants affected / at risk) | 0/2087 | 0/2368
Other Adverse Events (participants affected / at risk) | 0/2087 | 0/2368

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No